CLINICAL TRIAL: NCT04518358
Title: Expert Guiding Technology to Help Individuals With Developmental Challenges Build Life and Vocational Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John T. Nosek (Industry)
Responsible Party: Sponsor-Investigator, John T. Nosek, President & CEO, Guiding Technologies Corporation
Organization: Guiding Technologies Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R43MH121230-01 (NIH)
Record Dates: First submitted 2020-07-20; First posted 2020-08-19 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Autism Spectrum Disorder; Intellectual Disability
Keywords: expert software; behavioral intervention; Life Skill; Vocational Skill
MeSH Terms: conditions — Autism Spectrum Disorder; Intellectual Disability

STUDY DESIGN:
Intervention Model Description: A multiple probe design across participants will be used. This design necessitates a minimum of three participants to demonstrate experimental control, however 8 will be recruited. The small-N design yields much higher power and inferential validity than a traditional between-subject design, allowing for a much smaller n. The eight adults with ASD/ID will be divided into two groups, with four participants per group, which creates two sets of multiple probe designs. Baseline data will be collected for all participants (fidelity of treatment implementation for DSPs and independent completion of steps for adults with ASD/ID) for a minimum of three-to-five sessions prior to implementation of the intervention. Baseline data collection will continue until stability is achieved through each data point not exceeding 20% of mean responding during baseline. The intervention will be implemented in a staggered manner within each group in order to assess the effects of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of Expert Guiding Technology (Experimental)
  Interventions: Behavioral: Use of Expert Guiding Technology (GAINS) to Improve Live and Vocational Skills for Individuals with Developmental Challenges

INTERVENTIONS:
Behavioral: Use of Expert Guiding Technology (GAINS) to Improve Live and Vocational Skills for Individuals with Developmental Challenges — During the GAINS sessions, the Direct Support Professional (DSP) will follow the pre-programmed teaching protocol in the expert guiding technology. The system will provide step-by-step verbal prompts to the DSP throughout sessions. This includes which prompt to use for each step of the target skill, when to provide reinforcers, and which target task to work on. The system will also monitor the participant's (adults with ASD/ID) progress and notify the DSP if the target skill is mastered.

SUMMARY:
Clinical trials will evaluate the efficacy of expert guiding technology to support instructors to better help individuals with developmental challenges due to ASD and ID learn life and vocational skills. Single Case Research Designs (SCRD) will be used to evaluate expert guiding technology interventions to support Task Analysis. SCRDs are a viable alternative to large group studies such as randomized clinical trials. Single case studies involve repeated measures, and manipulation of an independent variable. SCRD studies allow for rigorous experimental evaluation of intervention effects and provide a strong basis for establishing causal inferences.

Research design: A multiple baseline across tasks or participants will be used to evaluate the impact of the expert guiding technology on staff and consumers' performance.

Dependent Variables. DV1: Staff performance: The percentage of teaching steps correctly implemented will be calculated and monitored. The teaching steps are predetermined including what types of prompts will be used for each step of the task analysis of the identified consumer's adaptive living skills, record data on consumer's performance, and the timing of delivery of reinforcers and prompts. DV2: Consumers' performance: The percentage of Independent completion of the steps of task analyses for identified daily living skills will be calculated and monitored. The completed step is considered "independent" when the consumer completed the step without prompts from the staff within five seconds of the initial instruction (discriminative stimulus) given or the completion of the previous step. DV3: Consumers' performance: the amount of time taken to independent completion.

Independent Variable: Versions of expert guiding technology to support instructors in providing Task Analyses instruction while collecting data on consumer performance.

GAINS: During the GAINS sessions, the staff will follow the pre-programmed teaching protocol in the expert guiding technology. The system will provide step-by-step verbal prompts to the staff throughout the sessions. This includes which prompt to use for each step, when to provide reinforcers, and which target task to work on. The system will also monitor the consumer's progress and notify the staff if the target task is mastered or not.

DETAILED DESCRIPTION:
Applied Behavior Analysis (ABA) remains the most effective and scientifically-validated approach to remediate the deficits caused by Autism Spectrum Disorders (ASD) and intellectual disabilities (ID). Clinical trials will evaluate the efficacy of expert guiding technology to support instructors to better help individuals with developmental challenges due to ASD and ID learn life and vocational skills. Single Case Research Designs (SCRD) will be used to evaluate expert guiding technology interventions to support Task Analysis. SCRDs are a viable alternative to large group studies such as randomized clinical trials. Single case studies involve repeated measures, and manipulation of an independent variable. SCRD studies allow for rigorous experimental evaluation of intervention effects and provide a strong basis for establishing causal inferences.

Research design: A multiple baseline across tasks or participants will be used to evaluate the impact of the expert guiding technology on staff and consumers' performance.

Dependent Variables. DV1: Staff performance: The percentage of teaching steps correctly implemented will be calculated and monitored. The teaching steps are predetermined including what types of prompts will be used for each step of the task analysis of the identified consumer's adaptive living skills, record data on consumer's performance, and the timing of delivery of reinforcers and prompts. DV2: Consumers' performance: The percentage of Independent completion of the steps of task analyses for identified daily living skills will be calculated and monitored. The completed step is considered "independent" when the consumer completed the step without prompts from the staff within five seconds of the initial instruction (discriminative stimulus) given or the completion of the previous step. DV3: Consumers' performance: the amount of time taken to independent completion.

Independent Variable: Versions of expert guiding technology to support instructors in providing Task Analyses instruction while collecting data on consumer performance.

GAINS: During the GAINS sessions, the staff will follow the pre-programmed teaching protocol in the expert guiding technology. The system will provide step-by-step verbal prompts to the staff throughout the sessions. This includes which prompt to use for each step, when to provide reinforcers, and which target task to work on. The system will also monitor the consumer's progress and notify the staff if the target task is mastered or not.

Procedural fidelity: procedural fidelity checklist will be implemented to ensure the accuracy of implementation of baseline and intervention procedures. The percentage of accurate implementation will be calculated by dividing the number of steps implemented accurately by the total steps of procedures multiplying by 100.

Develop and conduct survey of staff and consumers to evaluate social validity of expert guiding technology.

ELIGIBILITY:
Inclusion Criteria:

- Adults with Autism Spectrum Disorders and Intellectual Disabilities

Exclusion Criteria:

- none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John T Nosek, Ph.D., Principal Investigator — Guiding Technologies Corporation
Locations (1):
- Chimes Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
Any identifying information will be omitted from published or disseminated reports of the data to maintain confidentiality of subjects. Results of the study may be shared through conference presentations or written reports disseminated in peer-reviewed journals or other formats (e.gs., book chapters or grant proposals). In such cases, pseudonyms will be used and no identifying information (e.g., geographical location of subjects' residences) will be included when discussing results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available by the end of the project and for at least a year.
Access Criteria: Requests reviewed by the research team.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One adult participant with ASD took part in both SCED 1 and SCED 2. The enrollment number reflects the total unique number of participants.
Pre-assignment Details: Numbers in the table reflect dyads of instructor and adult with ASD.
Groups:
- Single Case Experimental Design (SCED) 1: Chimes staff identified the task of putting a computer shipping box together as very challenging. Consumers who could do this task were paid more for this task. This target task was observed and analyzed and nine task steps were identified. Because staff had identified this task as very challenging and since the steps to assemble the top were the same as assembling the bottom, the task was limited to assembling the bottom, then putting together the bottom with pre-assembled tops. The first SCED evaluated the efficacy of GAINS in helping to teach this task.
- Single Case Experimental Design (SCED) 2: Chimes staff identified the task of doing the laundry as a very useful and challenging task. This target task was observed and analyzed and 18 task steps were identified that required participants to complete tasks across a laundry room setup for training. 1) Pre-baseline DSP training: None. 2) Baseline: DSPs were given a list of the 18 task steps and told to teach as they normally would.
Period: Single Case Experimental Design (SCED) 1
Arm/Group | Single Case Experimental Design (SCED) 1 | Single Case Experimental Design (SCED) 2
Started (Each ARM consisted of 4 instructors and 4 adult participants with ASD.) | 4 | 0
Completed | 4 | 0
Not Completed | 0 | 0
Period: SCED 2
Arm/Group | Single Case Experimental Design (SCED) 1 | Single Case Experimental Design (SCED) 2
Started | 0 | 4
Completed | 0 | 4 (Four instructors completed the study and one initially enrolled instructor dropped out.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Separate baseline data were collected for instructors and adults with ASD.
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Case Experimental Design (SCED) 1 | Single Case Experimental Design (SCED) 2 | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants] — Population: Separate rows are used for instructors and adults with ASD.
  Participants
    SCED 1 Adults with ASD: number analyzed (Participants) | 4 | 0 | 4
    SCED 1 Adults with ASD: <=18 years | 0 |  | 0
    SCED 1 Adults with ASD: Between 18 and 65 years | 4 |  | 4
    SCED 1 Adults with ASD: >=65 years | 0 |  | 0
    SCED 2 Adults with ASD: number analyzed (Participants) | 0 | 4 | 4
    SCED 2 Adults with ASD: <=18 years | 0 | 0 | 0
    SCED 2 Adults with ASD: Between 18 and 65 years | 0 | 4 | 4
    SCED 2 Adults with ASD: >=65 years |  | 0 | 0
    SCED 1 + 2 Instructors: number analyzed (Participants) | 4 | 5 | 9
    SCED 1 + 2 Instructors: <=18 years | 0 | 0 | 0
    SCED 1 + 2 Instructors: Between 18 and 65 years | 4 | 5 | 9
    SCED 1 + 2 Instructors: >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Separate baseline data were collected for instructors and adults with ASD.
  Participants
    SCED 1 Adults with ASD: number analyzed (Participants) | 4 | 0 | 4
    SCED 1 Adults with ASD: Female | 0 |  | 0
    SCED 1 Adults with ASD: Male | 4 |  | 4
    SCED 2 Adults with ASD: number analyzed (Participants) | 0 | 4 | 4
    SCED 2 Adults with ASD: Female |  | 1 | 1
    SCED 2 Adults with ASD: Male |  | 3 | 3
    SCED 1 + 2 Instructors: number analyzed (Participants) | 4 | 5 | 9
    SCED 1 + 2 Instructors: Female | 2 | 4 | 6
    SCED 1 + 2 Instructors: Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Separate rows are used for instructors and adults with ASD.
  Participants
    SCED 1 Adults with ASD: number analyzed (Participants) | 4 | 0 | 4
    SCED 1 Adults with ASD: Hispanic or Latino | 0 |  | 0
    SCED 1 Adults with ASD: Not Hispanic or Latino | 4 |  | 4
    SCED 1 Adults with ASD: Unknown or Not Reported | 0 |  | 0
    SCED 2 Adults with ASD: number analyzed (Participants) | 0 | 4 | 4
    SCED 2 Adults with ASD: Hispanic or Latino |  | 0 | 0
    SCED 2 Adults with ASD: Not Hispanic or Latino |  | 4 | 4
    SCED 2 Adults with ASD: Unknown or Not Reported |  | 0 | 0
    SCED 1 + 2 Instructors: number analyzed (Participants) | 4 | 5 | 9
    SCED 1 + 2 Instructors: Hispanic or Latino | 0 | 1 | 1
    SCED 1 + 2 Instructors: Not Hispanic or Latino | 4 | 4 | 8
    SCED 1 + 2 Instructors: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: This measure is for instructors.
  participants
    United States: number analyzed (Participants) | 4 | 5 | 9
    United States | 4 | 5 | 9
Region of Enrollment [Number; unit: participants] — This measure is for SCED 1 Population: Separate rows are used for instructors and adults with ASD.
  participants
    United States: number analyzed (Participants) | 4 | 0 | 4
    United States | 4 |  | 4
Region of Enrollment [Number; unit: participants] — This measure is for SCED 2 Adults with ASD Population: Separate rows are used for instructors and adults with ASD.
  participants
    United States: number analyzed (Participants) | 0 | 4 | 4
    United States |  | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Fidelity of Treatment Implementation SCED 1 Dyad 1 Instructor
Description: One dependent measure is the fidelity of the teaching protocol implemented by DSPs. Each teaching protocol is comprised of a series of specific steps. Fidelity of the teaching protocol will be evaluated through collection of "yes" responses for accurately following the protocol and "no" responses for not accurately following the protocol for each step of the chain. The percentage of accurate implementation of the protocol will be calculated by dividing the steps marked with "yes" by the total number of the steps (sum of steps with "yes" and "no") and multiplied by 100. Data will be collected through multiple trials in order to perform visual analysis.
Time Frame: Single Case Research Design (SCRD): Multiple Baselines Repeated Measures Design. Repeated measures in baselines and repeated measures in the intervention will be taken after each intervention of the technology for approximately 3 weeks.
Population: Instructors within the first dyad.
Measure: Number; unit: Percent Correct
Groups:
- SCED 1 Instructor Dyad 1: Chimes staff identified the task of putting a computer shipping box together as very challenging. Consumers who could do this task were paid more for this task. This target task was observed and analyzed and nine task steps were identified.
Arm/Group | SCED 1 Instructor Dyad 1
Number analyzed (Participants) | 1
Percent Correct
  Session 1 - Baseline | 33
  Session 2 - Baseline | 11
  Session 3 - Baseline | 55
  Session 4 - Baseline | 55
  Session 5 - Baseline | 77
  Session 6 - Baseline | 66
  Session 7 - Intervention | 75
  Session 8 - Intervention | 100
  Session 9 - Intervention | 100
  Session 10 - Intervention | 100
  Session 11 - Intervention | 100
  Session 12 - Intervention | 100
  Session 13 - Intervention | 100
  Session 14 - Intervention | 100
  Session 15 - Intervention | 100
  Session 16 - Intervention | 100
  Session 17 - Intervention | 100
  Session 18 - Intervention | 100

2. Primary Outcome: Fidelity of Treatment Implementation SCED 1 Dyad 2 Instructor
Description: as for outcome 1
Time Frame: as for outcome 1
Population: SCED 1 Instructor in Dyad2
Measure: Number; unit: Percent Correct
Groups:
- SCED 1 Instructor Dyad 2: Chimes staff identified the task of putting a computer shipping box together as very challenging. Consumers who could do this task were paid more for this task. This target task was observed and analyzed and nine task steps were identified.
Arm/Group | SCED 1 Instructor Dyad 2
Number analyzed (Participants) | 1
Percent Correct
  Session 1 - Baseline | 33
  Session 2 - Baseline | 55
  Session 3 - Baseline | 100
  Session 4 - Intervention | 20
  Session 5 - Intervention | 86
  Session 6 - Intervention | 100
  Session 7 - Intervention | 100
  Session 8 - Intervention | 100
  Session 9 - Intervention | 100
  Session 10 - Intervention | 55
  Session 11 - Intervention | 77
  Session 12 - Intervention | 88
  Session 13 - Intervention | 100
  Session 14 - Intervention | 100
  Session 15 - Intervention | 100

3. Primary Outcome: Fidelity of Treatment Implementation SCED 1 Dyad 3 Instructor
Description: as for outcome 1
Time Frame: as for outcome 1
Population: SCED 1 Instructor in Dyad3
Measure: Number; unit: Percent Correct
Groups:
- SCED 1 Instructor Dyad 3: Chimes staff identified the task of putting a computer shipping box together as very challenging. Consumers who could do this task were paid more for this task. This target task was observed and analyzed and nine task steps were identified.
Arm/Group | SCED 1 Instructor Dyad 3
Number analyzed (Participants) | 1
Percent Correct
  Session 1 - Baseline | 100
  Session 2 - Baseline | 55
  Session 3 - Baseline | 44
  Session 4 - Baseline | 66
  Session 5 - Baseline | 88
  Session 6 - Baseline | 100
  Session 7 - Baseline | 77
  Session 8 - Baseline | 77
  Session 9 - Baseline | 88
  Session 10 - Intervention | 88
  Session 11 - Intervention | 88
  Session 12 - Intervention | 100
  Session 13 - Intervention | 100
  Session 14 - Intervention | 100
  Session 15 - Intervention | 100
  Session 16 - Intervention | 100
  Session 17 - Intervention | 100
  Session 18 - Intervention | 100
  Session 19 - Intervention | 100
  Session 20 - Intervention | 100
  Session 21 - Intervention | 100

4. Primary Outcome: Fidelity of Treatment Implementation SCED 1 Dyad 4 Instructor
Description: as for outcome 1
Time Frame: as for outcome 1
Population: SCED 1 Instructor in Dyad 4
Measure: Number; unit: Percent Correct
Groups:
- SCED 1 Instructor Dyad 4: Chimes staff identified the task of putting a computer shipping box together as very challenging. Consumers who could do this task were paid more for this task. This target task was observed and analyzed and nine task steps were identified.
Arm/Group | SCED 1 Instructor Dyad 4
Number analyzed (Participants) | 1
Percent Correct
  Session 1 - Baseline | 33
  Session 2 - Baseline | 55
  Session 3 - Baseline | 33
  Session 4 - Baseline | 33
  Session 5 - Baseline | 55
  Session 6 - Baseline | 88
  Session 7 - Baseline | 77
  Session 8 - Baseline | 88
  Session 9 - Baseline | 77
  Session 10 - Intervention | 100
  Session 11 - Intervention | 100
  Session 12 - Intervention | 88
  Session 13 - Intervention | 80
  Session 14 - Intervention | 88
  Session 15 - Intervention | 100
  Session 16 - Intervention | 100
  Session 17 - Intervention | 100
  Session 18 - Intervention | 100
  Session 19 - Intervention | 100
  Session 20 - Intervention | 100
  Session 21 - Intervention | 100

5. Primary Outcome: Fidelity of Treatment Implementation SCED 2 Dyad 1 Instructor
Description: as for outcome 1
Time Frame: as for outcome 1
Population: SCED 2 Instructor in Dyad 1
Measure: Number; unit: Percent Correct
Groups:
- SCED 2 Instructor Dyad 1: Chimes staff identified the task of doing the laundry as a very useful and challenging task. This target task was observed and analyzed and 18 task steps were identified that required participants to complete tasks across a laundry room setup for training. 1) Pre-baseline DSP training: None. 2) Baseline: DSPs were given a list of the 18 task steps and told to teach as they normally would.
Arm/Group | SCED 2 Instructor Dyad 1
Number analyzed (Participants) | 1
Percent Correct
  Session 1 - Baseline | 0
  Session 2 - Baseline | 5.56
  Session 3 - Baseline | 0
  Session 4 - Baseline | 0
  Session 5 - Intervention | 0
  Session 6 - Intervention | 88.89
  Session 7 - Intervention | 77.78
  Session 8 - Intervention | 72.22
  Session 9 - Intervention | 66.67
  Session 10 - Intervention | 83.33
  Session 11 - Intervention | 100
  Session 12 - Intervention | 88.89
  Session 13 - Intervention | 77.78
  Session 14 - Intervention | 61.11
  Session 15 - Intervention | 61.11
  Session 16 - Intervention | 83.33
  Session 17 - Intervention | 100
  Session 18 - Intervention | 100
  Session 19 - Intervention | 88.89
  Session 20 - Intervention | 100
  Session 21 - Intervention | 88.89
  Session 22 - Intervention | 100
  Session 23 - Intervention | 94.44
  Session 24 - Intervention | 94.44
  Session 25 - Intervention | 100
  Session 26 - Intervention | 83.33
  Session 27 - Intervention | 100
  Session 28 - Intervention | 72.22
  Session 29 - Intervention | 61.11
  Session 30 - Intervention | 77.78

6. Primary Outcome: Fidelity of Treatment Implementation SCED 2 Dyad 2 Instructor
Description: as for outcome 1
Time Frame: as for outcome 1
Population: SCED 2 Instructor in Dyad 2
Measure: Number; unit: Percent Correct
Groups:
- SCED 2 Instructor Dyad 2: Chimes staff identified the task of doing the laundry as a very useful and challenging task. This target task was observed and analyzed and 18 task steps were identified that required participants to complete tasks across a laundry room setup for training. 1) Pre-baseline DSP training: None. 2) Baseline: DSPs were given a list of the 18 task steps and told to teach as they normally would.
Arm/Group | SCED 2 Instructor Dyad 2
Number analyzed (Participants) | 1
Percent Correct
  Session 1 - Baseline | 0
  Session 2 - Baseline | 0
  Session 3 - Baseline | 0
  Session 4 - Baseline | 0
  Session 5 - Baseline | 0
  Session 6 - Baseline | 0
  Session 7 - Baseline | 0
  Session 8 - Baseline | 0
  Session 9 - Intervention | 77.78
  Session 10 - Intervention | 66.67
  Session 11 - Intervention | 100
  Session 12 - Intervention | 88.89
  Session 13 - Intervention | 88.89
  Session 14 - Intervention | 88.89
  Session 15 - Intervention | 100
  Session 16 - Intervention | 88.89
  Session 17 - Intervention | 88.89
  Session 18 - Intervention | 94.44
  Session 19 - Intervention | 100
  Session 20 - Intervention | 88.89
  Session 21 - Intervention | 88.89
  Session 22 - Intervention | 88.89
  Session 23 - Intervention | 100
  Session 24 - Intervention | 83.33
  Session 25 - Intervention | 100
  Session 26 - Intervention | 88.89

7. Primary Outcome: Fidelity of Treatment Implementation SCED 2 Dyad 3 Instructor
Description: as for outcome 1
Time Frame: as for outcome 1
Population: SCED 2 Instructor in Dyad 3
Measure: Number; unit: Percent Correct
Groups:
- SCED 2 Instructor Dyad 3: Chimes staff identified the task of doing the laundry as a very useful and challenging task. This target task was observed and analyzed and 18 task steps were identified that required participants to complete tasks across a laundry room setup for training. 1) Pre-baseline DSP training: None. 2) Baseline: DSPs were given a list of the 18 task steps and told to teach as they normally would.
Arm/Group | SCED 2 Instructor Dyad 3
Number analyzed (Participants) | 1
Percent Correct
  Session 1 - Baseline | 0
  Session 2 - Baseline | 0
  Session 3 - Baseline | 0
  Session 4 - Baseline | 0
  Session 5 - Baseline | 0
  Session 6 - Baseline | 11.11
  Session 7 - Baseline | 11.11
  Session 8 - Baseline | 0
  Session 9 - Baseline | 0
  Session 10 - Baseline | 0
  Session 11 - Baseline | 0
  Session 12 - Baseline | 0
  Session 13 - Intervention | 94.44
  Session 14 - Intervention | 83.33
  Session 15 - Intervention | 100
  Session 16 - Intervention | 100
  Session 17 - Intervention | 94.44
  Session 18 - Intervention | 100
  Session 19 - Intervention | 94.44
  Session 20 - Intervention | 100
  Session 21 - Intervention | 88.89
  Session 22 - Intervention | 94.44
  Session 23 - Intervention | 94.44
  Session 24 - Intervention | 88.89
  Session 25 - Intervention | 100
  Session 26 - Intervention | 94.44
  Session 27 - Intervention | 88.89
  Session 28 - Intervention | 88.89
  Session 29 - Intervention | 88.89
  Session 30 - Intervention | 83.33

8. Primary Outcome: Fidelity of Treatment Implementation SCED 2 Dyad 4 Instructor
Description: as for outcome 1
Time Frame: as for outcome 1
Population: SCED 2 Instructor in Dyad 4
Measure: Number; unit: Percent Correct
Groups:
- SCED 2 Instructor Dyad 4: Chimes staff identified the task of doing the laundry as a very useful and challenging task. This target task was observed and analyzed and 18 task steps were identified that required participants to complete tasks across a laundry room setup for training. 1) Pre-baseline DSP training: None. 2) Baseline: DSPs were given a list of the 18 task steps and told to teach as they normally would.
Arm/Group | SCED 2 Instructor Dyad 4
Number analyzed (Participants) | 1
Percent Correct
  Session 1 - Baseline | 0
  Session 2 - Baseline | 0
  Session 3 - Baseline | 0
  Session 4 - Baseline | 0
  Session 5 - Baseline | 0
  Session 6 - Baseline | 0
  Session 7 - Baseline | 22.22
  Session 8 - Baseline | 0
  Session 9 - Baseline | 0
  Session 10 - Baseline | 0
  Session 11 - Baseline | 0
  Session 12 - Baseline | 11.11
  Session 13 - Baseline | 5.56
  Session 14 - Baseline | 33.33
  Session 15 - Baseline | 27.78
  Session 16 - Baseline | 11.11
  Session 17 - Intervention | 94.44
  Session 18 - Intervention | 88.89
  Session 19 - Intervention | 94.44
  Session 20 - Intervention | 83.33
  Session 21 - Intervention | 77.78
  Session 22 - Intervention | 88.89

9. Primary Outcome: Independent Completion of Steps SCED 1 Dyad 1 Adult With ASD
Description: Each target skill performed by adults with ASD/ID will be task analyzed. Tasks analysis involves breaking the skill down into smaller steps. The percentage of independent completion of steps will be calculated by dividing the number of independently completed steps by the total number of steps and multiplying by 100. Data will be captured through multiple trials to make visual analysis possible.
Time Frame: as for outcome 1
Population: SCED 1 Dyad 1 Adult with ASD
Measure: Number; unit: Percent Correct
Groups:
- SCED 1 Dyad 1 Adult With ASD: Chimes staff identified the task of putting a computer shipping box together as very challenging. Consumers who could do this task were paid more for this task. This target task was observed and analyzed and nine task steps were identified.
Arm/Group | SCED 1 Dyad 1 Adult With ASD
Number analyzed (Participants) | 1
Percent Correct
  Session 1 - Baseline | 22
  Session 2 - Baseline | 33
  Session 3 - Baseline | 55
  Session 4 - Baseline | 44
  Session 5 - Baseline | 77
  Session 6 - Baseline | 77
  Session 7 - Intervention | 33
  Session 8 - Intervention | 77
  Session 9 - Intervention | 88
  Session 10 - Intervention | 77
  Session 11 - Intervention | 88
  Session 12 - Intervention | 77
  Session 13 - Intervention | 66
  Session 14 - Intervention | 77
  Session 15 - Intervention | 88
  Session 16 - Intervention | 55
  Session 17 - Intervention | 77
  Session 18 - Intervention | 77

10. Primary Outcome: Independent Completion of Steps SCED 1 Dyad 2 Adult With ASD
Description: as for outcome 9
Time Frame: as for outcome 1
Population: SCED 1 Dyad 2 Adult with ASD
Measure: Number; unit: Percent Correct
Groups:
- SCED 1 Dyad 2 Adult With ASD: Chimes staff identified the task of putting a computer shipping box together as very challenging. Consumers who could do this task were paid more for this task. This target task was observed and analyzed and nine task steps were identified.
Arm/Group | SCED 1 Dyad 2 Adult With ASD
Number analyzed (Participants) | 1
Percent Correct
  Session 1 - Baseline | 22
  Session 2 - Baseline | 44
  Session 3 - Baseline | 55
  Session 4 - Intervention | 80
  Session 5 - Intervention | 66
  Session 6 - Intervention | 66
  Session 7 - Intervention | 77
  Session 8 - Intervention | 66
  Session 9 - Intervention | 88
  Session 10 - Intervention | 55
  Session 11 - Intervention | 77
  Session 12 - Intervention | 88
  Session 13 - Intervention | 77
  Session 14 - Intervention | 100
  Session 15 - Intervention | 88

11. Primary Outcome: Independent Completion of Steps SCED 1 Dyad 3 Adult With ASD
Description: as for outcome 9
Time Frame: as for outcome 1
Population: SCED 1 Dyad 3 Adult with ASD
Measure: Number; unit: Percent Correct
Groups:
- SCED 1 Dyad 3 Adult With ASD: Chimes staff identified the task of putting a computer shipping box together as very challenging. Consumers who could do this task were paid more for this task. This target task was observed and analyzed and nine task steps were identified.
Arm/Group | SCED 1 Dyad 3 Adult With ASD
Number analyzed (Participants) | 1
Percent Correct
  Session 1 - Baseline | 66
  Session 2 - Baseline | 77
  Session 3 - Baseline | 33
  Session 4 - Baseline | 33
  Session 5 - Baseline | 66
  Session 6 - Baseline | 100
  Session 7 - Baseline | 88
  Session 8 - Baseline | 77
  Session 9 - Baseline | 100
  Session 10 - Intervention | 66
  Session 11 - Intervention | 88
  Session 12 - Intervention | 88
  Session 13 - Intervention | 88
  Session 14 - Intervention | 88
  Session 15 - Intervention | 100
  Session 16 - Intervention | 100
  Session 17 - Intervention | 100
  Session 18 - Intervention | 100
  Session 19 - Intervention | 100
  Session 20 - Intervention | 100
  Session 21 - Intervention | 100

12. Primary Outcome: Independent Completion of Steps SCED 1 Dyad 4 Adult With ASD
Description: as for outcome 9
Time Frame: as for outcome 1
Population: SCED 1 Dyad 4 Adult with ASD
Measure: Number; unit: Percent Correct
Groups:
- SCED 1 Dyad 4 Adult With ASD: Chimes staff identified the task of putting a computer shipping box together as very challenging. Consumers who could do this task were paid more for this task. This target task was observed and analyzed and nine task steps were identified.
Arm/Group | SCED 1 Dyad 4 Adult With ASD
Number analyzed (Participants) | 1
Percent Correct
  Session 1 - Baseline | 33
  Session 2 - Baseline | 55
  Session 3 - Baseline | 55
  Session 4 - Baseline | 44
  Session 5 - Baseline | 55
  Session 6 - Baseline | 77
  Session 7 - Baseline | 77
  Session 8 - Baseline | 55
  Session 9 - Baseline | 77
  Session 10 - Intervention | 86
  Session 11 - Intervention | 66
  Session 12 - Intervention | 100
  Session 13 - Intervention | 75
  Session 14 - Intervention | 77
  Session 15 - Intervention | 75
  Session 16 - Intervention | 88
  Session 17 - Intervention | 88
  Session 18 - Intervention | 77
  Session 19 - Intervention | 100
  Session 20 - Intervention | 100
  Session 21 - Intervention | 100

13. Primary Outcome: Independent Completion of Steps SCED 2 Dyad 1 Adult With ASD
Description: as for outcome 9
Time Frame: as for outcome 1
Population: SCED 2 Dyad 1 Adult with ASD
Measure: Number; unit: Percent Correct
Groups:
- SCED 2 Dyad 1 Adult With ASD: Chimes staff identified the task of doing the laundry as a very useful and challenging task. This target task was observed and analyzed and 18 task steps were identified that required participants to complete tasks across a laundry room setup for training. 1) Pre-baseline DSP training: None. 2) Baseline: DSPs were given a list of the 18 task steps and told to teach as they normally would.
Arm/Group | SCED 2 Dyad 1 Adult With ASD
Number analyzed (Participants) | 1
Percent Correct
  Session 1 - Baseline | 0
  Session 2 - Baseline | 5.56
  Session 3 - Baseline | 0
  Session 4 - Baseline | 0
  Session 5 - Intervention | 0
  Session 6 - Intervention | 50
  Session 7 - Intervention | 38.89
  Session 8 - Intervention | 44.44
  Session 9 - Intervention | 55.56
  Session 10 - Intervention | 50
  Session 11 - Intervention | 66.67
  Session 12 - Intervention | 44.44
  Session 13 - Intervention | 50
  Session 14 - Intervention | 27.78
  Session 15 - Intervention | 66.67
  Session 16 - Intervention | 50.00
  Session 17 - Intervention | 72.22
  Session 18 - Intervention | 66.67
  Session 19 - Intervention | 77.78
  Session 20 - Intervention | 72.22
  Session 21 - Intervention | 72.22
  Session 22 - Intervention | 38.89
  Session 23 - Intervention | 61.11
  Session 24 - Intervention | 61.11
  Session 25 - Intervention | 72.22
  Session 26 - Intervention | 44.44
  Session 27 - Intervention | 77.78
  Session 28 - Intervention | 55.56
  Session 29 - Intervention | 61.11
  Session 30 - Intervention | 66.67

14. Primary Outcome: Independent Completion of Steps SCED 2 Dyad 2 Adult With ASD
Description: as for outcome 9
Time Frame: as for outcome 1
Population: SCED 2 Dyad 2 Adult with ASD
Measure: Number; unit: Percent Correct
Groups:
- SCED 2 Dyad 2 Adult With ASD: Chimes staff identified the task of doing the laundry as a very useful and challenging task. This target task was observed and analyzed and 18 task steps were identified that required participants to complete tasks across a laundry room setup for training. 1) Pre-baseline DSP training: None. 2) Baseline: DSPs were given a list of the 18 task steps and told to teach as they normally would.
Arm/Group | SCED 2 Dyad 2 Adult With ASD
Number analyzed (Participants) | 1
Percent Correct
  Session 1 - Baseline | 0
  Session 2 - Baseline | 0
  Session 3 - Baseline | 0
  Session 4 - Baseline | 11.11
  Session 5 - Baseline | 0
  Session 6 - Baseline | 16.67
  Session 7 - Baseline | 11.11
  Session 8 - Baseline | 0
  Session 9 - Intervention | 50
  Session 10 - Intervention | 38.89
  Session 11 - Intervention | 88.89
  Session 12 - Intervention | 11.11
  Session 13 - Intervention | 22.22
  Session 14 - Intervention | 55.56
  Session 15 - Intervention | 44.44
  Session 16 - Intervention | 61.11
  Session 17 - Intervention | 50
  Session 18 - Intervention | 66.67
  Session 19 - Intervention | 83.33
  Session 20 - Intervention | 55.56
  Session 21 - Intervention | 50
  Session 22 - Intervention | 55.56
  Session 23 - Intervention | 66.67
  Session 24 - Intervention | 50
  Session 25 - Intervention | 50
  Session 26 - Intervention | 72.22

15. Primary Outcome: Independent Completion of Steps SCED 2 Dyad 3 Adult With ASD
Description: as for outcome 9
Time Frame: as for outcome 1
Population: SCED 2 Dyad 3 Adult with ASD
Measure: Number; unit: Percent Correct
Groups:
- SCED 2 Dyad 3 Adult With ASD: Chimes staff identified the task of doing the laundry as a very useful and challenging task. This target task was observed and analyzed and 18 task steps were identified that required participants to complete tasks across a laundry room setup for training. 1) Pre-baseline DSP training: None. 2) Baseline: DSPs were given a list of the 18 task steps and told to teach as they normally would.
Arm/Group | SCED 2 Dyad 3 Adult With ASD
Number analyzed (Participants) | 1
Percent Correct
  Session 1 - Baseline | 0
  Session 2 - Baseline | 0
  Session 3 - Baseline | 0
  Session 4 - Baseline | 0
  Session 5 - Baseline | 0
  Session 6 - Baseline | 0
  Session 7 - Baseline | 5.56
  Session 8 - Baseline | 0
  Session 9 - Baseline | 0
  Session 10 - Baseline | 5.56
  Session 11 - Baseline | 0
  Session 12 - Baseline | 0
  Session 13 - Intervention | 0
  Session 14 - Intervention | 0
  Session 15 - Intervention | 11.11
  Session 16 - Intervention | 22.22
  Session 17 - Intervention | 5.56
  Session 18 - Intervention | 27.78
  Session 19 - Intervention | 5.56
  Session 20 - Intervention | 16.67
  Session 21 - Intervention | 22.22
  Session 22 - Intervention | 11.11
  Session 23 - Intervention | 38.89
  Session 24 - Intervention | 44.44
  Session 25 - Intervention | 55.56
  Session 26 - Intervention | 33.33
  Session 27 - Intervention | 38.89
  Session 28 - Intervention | 66.67
  Session 29 - Intervention | 38.89
  Session 30 - Intervention | 33.33

16. Primary Outcome: Independent Completion of Steps SCED 2 Dyad 4 Adult With ASD
Description: as for outcome 9
Time Frame: as for outcome 1
Population: SCED 2 Dyad 4 Adult with ASD
Measure: Number; unit: Percent Correct
Groups:
- SCED 2 Dyad 4 Adult With ASD: Chimes staff identified the task of doing the laundry as a very useful and challenging task. This target task was observed and analyzed and 18 task steps were identified that required participants to complete tasks across a laundry room setup for training. 1) Pre-baseline DSP training: None. 2) Baseline: DSPs were given a list of the 18 task steps and told to teach as they normally would.
Arm/Group | SCED 2 Dyad 4 Adult With ASD
Number analyzed (Participants) | 1
Percent Correct
  Session 1 - Baseline | 0
  Session 2 - Baseline | 0
  Session 3 - Baseline | 0
  Session 4 - Baseline | 0
  Session 5 - Baseline | 0
  Session 6 - Baseline | 0
  Session 7 - Baseline | 22.22
  Session 8 - Baseline | 0
  Session 9 - Baseline | 0
  Session 10 - Baseline | 0
  Session 11 - Baseline | 0
  Session 12 - Baseline | 11.11
  Session 13 - Baseline | 5.56
  Session 14 - Baseline | 33.33
  Session 15 - Baseline | 27.78
  Session 16 - Baseline | 11.11
  Session 17 - Intervention | 72.22
  Session 18 - Intervention | 61.11
  Session 19 - Intervention | 94.44
  Session 20 - Intervention | 72.22
  Session 21 - Intervention | 38.89
  Session 22 - Intervention | 83.33

17. Secondary Outcome: Number of Sessions to Skill Acquisition SCED 1 Dyad 3 Adult With ASD
Description: In addition to the level of independence of adults with ASD/ID, the number of sessions required for them to acquire the target skill will be monitored. The criterion of skill acquisition is 90% or above of independent completion of steps for three consecutive sessions.
Time Frame: Single Case Research Design (SCRD): Multiple Baselines Repeated Measures Design. Repeated measures in baselines and repeated measures in the intervention will be taken after each intervention of the technology for approximately 3 weeks. There will be two
Population: SCED 1 Dyad 3 Adult with ASD
Measure: Number; unit: Number of Sessions to reach independence
Arm/Group | SCED 1 Dyad 3 Adult With ASD
Number analyzed (Participants) | 1
Number of Sessions to reach independence | 17

18. Secondary Outcome: Number of Sessions to Skill Acquisition SCED 1 Dyad 4 Adult With ASD
Description: as for outcome 17
Time Frame: as for outcome 17
Population: SCED 1 Dyad 4 Adult with ASD
Measure: Number; unit: Number of Sessions to reach independence
Arm/Group | SCED 1 Dyad 4 Adult With ASD
Number analyzed (Participants) | 1
Number of Sessions to reach independence | 21

ADVERSE EVENTS:
Description: Exempt protocol, teaching under typical conditions. All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Evaluation of Expert Guiding Technology
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT04518358/Prot_000.pdf